CLINICAL TRIAL: NCT04793217
Title: Project Someleze: A Randomized Trial of ImpACT+, a Coping Intervention to Improve Clinical and Mental Health Outcomes Among HIV-infected Women With Sexual Trauma in South Africa
Brief Title: A Randomized Trial of ImpACT+, a Coping Intervention for HIV Infected Women With Sexual Trauma in South Africa
Acronym: ImpACT+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Cape Town (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathleen J. Sikkema, PhD, Stephen Smith Professor of Sociomedical Sciences; Chair, Department of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAS3667; 1R01MH118004 (NIH)
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HIV; Trauma Exposure
Keywords: South Africa; HIV; Mental health; Trauma; Women
MeSH Terms: conditions — Psychological Well-Being; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Improving AIDS Care after Trauma+ (Experimental): ImpACT+ (Improving AIDS Care after Trauma+), is an individual-level coping intervention to address traumatic stress and HIV care engagement among South African women with sexual trauma histories. The ImpACT+ individual sessions will focus on coping skills and care engagement during an early critical period, while maintenance check-ins will serve to reinforce positive change and support the ongoing implementation of skills as new challenges arise.
  Interventions: Behavioral: Improving AIDS Care After Trauma +
- Adapted Problem-Solving Therapy (Active Comparator): Participants randomly assigned to the control condition will receive a brief adapted version of problem-solving therapy (PST), based on Problem Management Plus, a component of the World Health Organization (WHO) Mental Health Gap Action Programme (mhGAP). PST is a psychoeducational treatment focused on managing the negative effects of stressful life events. PST has been found to be effective for a range of problems, such as depression, and is recommended for implementation in low-resource settings.
  Interventions: Behavioral: Adapted Problem-Solving Therapy

INTERVENTIONS:
Behavioral: Improving AIDS Care After Trauma + — ImpACT+ integrates skills for HIV treatment adherence and coping with trauma, tailored to the South African context. This includes exploration of values informing care engagement, recognizing the synergistic stress of sexual trauma and HIV, understanding the contribution of stressors to maladaptive coping, and developing adaptive methods for coping as alternatives to avoidance. ImpACT+ will be delivered in private spaces at the primary care clinic and will consist of 6 individual sessions followed by 6 maintenance check-ins. Individual sessions focus on coping, adherence, and care engagement during an early critical period, while maintenance check-ins reinforce positive change and support ongoing implementation of skills. Evidence supports a 6-session format in low-resource settings. Individual sessions will begin within 2 weeks after the baseline survey and be completed by the 4-month assessment. Maintenance check-ins will begin following the 4-month assessment.
  Arms: Improving AIDS Care after Trauma+
Behavioral: Adapted Problem-Solving Therapy — Participants will receive three weekly individual sessions of adapted PST. The goal of PST is to identify problems that interfere with daily activities and address them through problem-orientation work. We anticipate stressors will include (a) relationship difficulties, including family stress, (b) financial stress and unemployment, (c) general impact of HIV infection, and (d) overall chronic stress. Thus, PST may indirectly address stressors that may impact care engagement, but will not address the intersection of HIV and trauma specifically.
  Arms: Adapted Problem-Solving Therapy

SUMMARY:
ImpACT+ (Improving AIDS Care after Trauma+), is an individual-level coping intervention to address traumatic stress and HIV care engagement among South African women with sexual trauma histories. We propose a full-scale randomized controlled trial to examine the effect of ImpACT+ on clinical outcomes in the period after ART initiation and to understand mental health and behavioral mechanisms through which viral suppression can be achieved. ImpACT+ will target women who are initiating ART in order to take advantage of a window of opportunity in HIV care and maximize care engagement. The aims are to test the effectiveness of ImpACT+ and explore its potential for implementation.

DETAILED DESCRIPTION:
Addressing sexual trauma in the context of HIV care is essential to improve clinical outcomes and mental health among women in South Africa. Women represent nearly two-thirds of the South African HIV epidemic, and they report disproportionately high rates of sexual trauma, which negatively impacts their mental health and may lead to avoidant coping behaviors. The psychological sequaelae of trauma can adversely impact retention in HIV care and adherence to antiretroviral therapy (ART), which may in turn reduce viral suppression and increase the risk of HIV transmission to others. HIV care engagement may be particularly challenging in South Africa, where women face dual epidemics of HIV and sexual violence, with limited access to mental health treatment. In this setting, interventions that address barriers to effective HIV care engagement and improve health outcomes across the care continuum are urgently needed. The primary objective of this study is to evaluate the effectiveness of ImpACT+ (Improving AIDS Care after Trauma+), an individual-level intervention based on theories of stress and coping, on clinical outcomes among HIV-infected women with sexual trauma. Secondary objectives include determining whether reductions in traumatic stress and avoidant coping mediate intervention effects on clinical outcomes, and assessing potential for scalability and full-scale implementation. ImpACT+ was developed and culturally adapted to the South African context, targeting women who are initiating ART (classified clinically as naïve initiators, restarters or defaulters) to make use of a window of opportunity in HIV care and maximize impact on care engagement. The proposed five-year study seeks to rigorously evaluate ImpACT+, using a hybrid effectiveness-implementation design (Hybrid Type I), with three specific aims: (1) evaluate the effectiveness of ImpACT+ on viral suppression, ART adherence, and HIV care engagement; (2) assess the degree to which reductions in PTSD symptoms and avoidant coping mediate intervention effects; and (3) explore potential for scalability and full-scale implementation. The trial will enroll 350 women who have initiated ART and have a history of sexual trauma and elevated traumatic stress. Participants will be randomized to the ImpACT+ intervention condition (six weekly sessions, with six maintenance check-ins over the 12-month follow-up period) or the control condition (three weekly sessions of Problem Solving Therapy (PST)). All participants will complete a baseline assessment at enrollment (within four months of initiating ART), with additional behavioral assessments and viral load testing at 4-month, 8-month, and 12-month follow-up. ART adherence will also be assessed using dried blood spot (DBS) biomarkers, and care engagement data will be extracted from medical records at the end of the study period. This study is one of the first full-scale trials of a trauma-informed intervention on clinical outcomes for HIV-infected women. If effective, ImpACT+ will fill a critical void in evidence-based trauma interventions in this setting and combat the drop-off across the HIV continuum of care in South Africa, as well as inform such approaches in the U.S. and globally.

ELIGIBILITY:
Inclusion Criteria:

* Women with HIV who receive care at either study clinic
* >2 weeks to <4 months since ART initiation
* History of sexual trauma
* Meets criteria for traumatic stress
* Xhosa speaking

Exclusion Criteria:

- High suicide risk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women are eligible for this study
Enrollment: 350 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Viral suppression/viral load | Up to 12 months
  HIV-1 RNA viral load (COBAS AmpliPrep/COBAS TaqMan HIV-1 Test, v2.0, Roche). Viral suppression defined as <50 copies/ml. Continuous measures of viral load, modeled using a log10 transformation.

SECONDARY OUTCOMES:
HIV Care Engagement- Number of Missed Visits | Up to 12 months
  The number of missed visits as determined by medical record review.
HIV Care Engagement- Visit Adherence | Up to 12 months
  Visit adherence defined as the number of scheduled visits attended.
HIV Care Engagement- Gaps in Care | Up to 12 months
  Gaps in care defined as whether >90 days have elapse between visits, as determined by medical record abstraction.
HIV Care Engagement- Visit Constancy | Up to 12 months
  Visit constancy defined as the number of 90-day intervals with >1 completed visit, determined by medical record abstraction.
ART Adherence - Dried Blood Spots | Up to 12 months
  Dried blood spots measuring levels of tenofovir-diphosphate, dichotomized as adherent or non-adherent.
ART Adherence - Pharmacy Visits | Up to 12 months
  ART adherence as defined by the number of pharmacy visits. Determined through medical record abstraction.
ART Adherence - Pharmacy Refill | Up to 12 months
  ART adherence as defined by pharmacy refill data. Determined through medical record abstraction.

OTHER OUTCOMES:
Coping Strategies Scale Score | Up to 12 months
  Self report, measured by Coping Strategies scale (Sikkema et al., 2018; based on Carver, 1997; Folkman & Lazarus, 1988; Hansen et al., 2013; Namir et al., 1987). Coping will be assessed using 41 items that were previously used to measure coping in Sub-Saharan Africa or among HIV-infected individuals. Participants will be asked how often they used these strategies in the past month to help deal with their HIV illness (1 = not at all to 4 = most of the time).
Traumatic Stress Score | Up to 12 months
  Self report, measured by PTSD Checklist-Civilian version for the The Diagnostic and Statistical Manual of Mental Disorders (DSM-5; Blevins CA, Weathers FW, Davis MT, Witte TK, and Domino JKL, 2015). PCL-5 [51], a 20-item self-report questionnaire, will assess severity of symptoms that parallel DSM-5 diagnostic criteria for PTSD. Participants will be asked to indicate the extent to which they were bothered by problems experienced in the past month in relation to a traumatic experience of abuse or act of violence (0 = not at all to 4 = extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen J Sikkema, PhD, Principal Investigator — Columbia University
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share an anonymized dataset following publications.
Supporting Information: Study Protocol, SAP
Time Frame: Following outcome publications.
Access Criteria: Access will be granted upon reasonable requests.

REFERENCES:
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Folkman S, Lazarus RS. The relationship between coping and emotion: implications for theory and research. Soc Sci Med. 1988;26(3):309-17. doi: 10.1016/0277-9536(88)90395-4. PMID 3279520
- [Background] Hansen NB, Harrison B, Fambro S, Bodnar S, Heckman TG, Sikkema KJ. The structure of coping among older adults living with HIV/AIDS and depressive symptoms. J Health Psychol. 2013 Feb;18(2):198-211. doi: 10.1177/1359105312440299. Epub 2012 Mar 27. PMID 22453164
- [Background] Knettel BA, Robertson C, Ciya N, Coleman JN, Elliott SA, Joska JA, Sikkema KJ. "I cannot change what happened to me, but I can learn to change how I feel": A case study from ImpACT, an intervention for women with a history of sexual trauma who are living with HIV in Cape Town, South Africa. Psychotherapy (Chic). 2020 Mar;57(1):90-96. doi: 10.1037/pst0000263. Epub 2019 Dec 19. PMID 31855042
- [Background] Knettel BA, Mulawa MI, Knippler ET, Ciya N, Robertson C, Joska JA, Sikkema KJ. Women's perspectives on ImpACT: a coping intervention to address sexual trauma and improve HIV care engagement in Cape Town, South Africa. AIDS Care. 2019 Nov;31(11):1389-1396. doi: 10.1080/09540121.2019.1587368. Epub 2019 Mar 1. PMID 30821168
- [Background] Meade CS, Kershaw TS, Hansen NB, Sikkema KJ. Long-term correlates of childhood abuse among adults with severe mental illness: adult victimization, substance abuse, and HIV sexual risk behavior. AIDS Behav. 2009 Apr;13(2):207-16. doi: 10.1007/s10461-007-9326-4. Epub 2007 Oct 30. PMID 17968646
- [Background] Namir S, Wolcott DL, Fawzy FI, Alumbaugh MJ. Coping with AIDS: Psychological and health implications. J Appl Soc Psychol. 1987;17(3):309-328. doi:10.1111/j.1559-1816.1987.tb00316.x
- [Background] Sikkema KJ, Choi KW, Robertson C, Knettel BA, Ciya N, Knippler ET, Watt MH, Joska JA. Development of a coping intervention to improve traumatic stress and HIV care engagement among South African women with sexual trauma histories. Eval Program Plann. 2018 Jun;68:148-156. doi: 10.1016/j.evalprogplan.2018.02.007. Epub 2018 Mar 6. PMID 29597104
- [Background] Sikkema KJ, Mulawa MI, Robertson C, Watt MH, Ciya N, Stein DJ, Cherenack EM, Choi KW, Kombora M, Joska JA. Improving AIDS Care After Trauma (ImpACT): Pilot Outcomes of a Coping intervention Among HIV-Infected Women with Sexual Trauma in South Africa. AIDS Behav. 2018 Mar;22(3):1039-1052. doi: 10.1007/s10461-017-2013-1. PMID 29270789
- [Background] Sikkema KJ, Ranby KW, Meade CS, Hansen NB, Wilson PA, Kochman A. Reductions in traumatic stress following a coping intervention were mediated by decreases in avoidant coping for people living with HIV/AIDS and childhood sexual abuse. J Consult Clin Psychol. 2013 Apr;81(2):274-83. doi: 10.1037/a0030144. Epub 2012 Oct 1. PMID 23025248
- [Background] Sikkema KJ, Wilson PA, Hansen NB, Kochman A, Neufeld S, Ghebremichael MS, Kershaw T. Effects of a coping intervention on transmission risk behavior among people living with HIV/AIDS and a history of childhood sexual abuse. J Acquir Immune Defic Syndr. 2008 Apr 1;47(4):506-13. doi: 10.1097/QAI.0b013e318160d727. PMID 18176319
- [Background] Watt MH, Dennis AC, Choi KW, Ciya N, Joska JA, Robertson C, Sikkema KJ. Impact of Sexual Trauma on HIV Care Engagement: Perspectives of Female Patients with Trauma Histories in Cape Town, South Africa. AIDS Behav. 2017 Nov;21(11):3209-3218. doi: 10.1007/s10461-016-1617-1. PMID 27866288
- [Derived] Rabie S, Poudyal A, Mirti A, Wilson P, Joska JA, Sikkema KJ. The Factorial Structure, Reliability, and Validity of a Coping Measure Among Women with HIV and Sexual Trauma in Cape Town, South Africa. AIDS Behav. 2025 Sep 23. doi: 10.1007/s10461-025-04886-6. Online ahead of print. PMID 40983787
- [Derived] Sikkema KJ, Rabie S, King A, Watt MH, Mulawa MI, Andersen LS, Wilson PA, Marais A, Ndwandwa E, Majokweni S, Orrell C, Joska JA. ImpACT+, a coping intervention to improve clinical outcomes for women living with HIV and sexual trauma in South Africa: study protocol for a randomized controlled trial. Trials. 2022 Aug 18;23(1):680. doi: 10.1186/s13063-022-06655-5. PMID 35982485